CLINICAL TRIAL: NCT01450280
Title: A Phase Ia Study to Assess the Safety and Immunogenicity of New Malaria Vaccine Candidates ChAd63 CS Administered Alone and With MVA CS
Brief Title: Safety and Immunogenicity of New Malaria Vaccine Candidate ChAd63 CS Administered Alone and With MVA CS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC038
Record Dates: First submitted 2011-10-03; First posted 2011-10-12 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1A (Experimental): AdCh63 CS 5x10^9 vp
  Interventions: Biological: ChAd63 CS
- Group 1B (Experimental): ChAd63 CS 5x10^9 vp Day 0; MVA CS 2x10^8 pfu Day 56
  Interventions: Biological: ChAd63 CS, MVA CS
- Group 2A (Experimental): AdCh63 CS 5 x 10^10 vp
  Interventions: Biological: ChAd63 CS
- Group 2B (Experimental): ChAd63 CS 5x10^10 vp Day 0; MVA CS 2x10^8 pfu Day 56
  Interventions: Biological: ChAd63, MVA CS

INTERVENTIONS:
Biological: ChAd63 CS — ChAd63 CS 5x10^9 vp intra-muscularly Day 0
  Arms: Group 1A
Biological: ChAd63 CS, MVA CS — ChAd63 CS 5x10^9 vp intra-muscularly Day 0; MVA CS 2x10^8 pfu intra-muscularly Day 56
  Arms: Group 1B
Biological: ChAd63 CS — ChAd63 CS 5x10^10 vp intra-muscularly Day 0
  Arms: Group 2A
Biological: ChAd63, MVA CS — ChAd63 CS 5x10^10 vp intra-muscularly Day 0; MVA CS 2x10^8 pfu intra-muscularly Day 56
  Arms: Group 2B

SUMMARY:
This is an open label phase I study, to assess the safety of a novel malaria vaccine, AdCh63 CS, simian adenovirus encoding Plasmodium falciparum liver stage antigen, Circumsporozoite protein. All volunteers recruited will be healthy adults. They will be primed with various doses of AdCh63 CS administered intramuscularly. Some of the volunteers will receive a booster vaccination with MVA CS administered via intramuscular route. Safety data will be collected for each vaccination regimen. Secondary aim of this study will be to assess the immune responses generated by vaccination.

ELIGIBILITY:
Inclusion Criteria

* Healthy adults aged 18 to 50 years
* Able and willing (in the Investigator"s opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer"s medical history with their General Practitioner
* Women only: Must practice continuous effective contraception for the duration of the study
* Agreement to refrain from blood donation during the course of the study and for 6 months after the end of their involvement in the study.
* Written informed consent

Exclusion Criteria:

* History of clinical P. falciparum malaria
* Travel to a malaria endemic region during the study period or within the preceding six months with a significant risk of malaria exposure.
* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period.
* Prior receipt of an investigational malaria vaccine or any other investigational vaccine likely to impact on interpretation of the trial data.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* Pregnancy, breast feeding or intention to become pregnant during the study
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine e.g. egg products, Kathon.
* History of clinically significant contact dermatitis.
* Any history of anaphylaxis post vaccination.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study.
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Seropositive for hepatitis B surface antigen (HBsAg).
* Seropositive for hepatitis C virus (antibodies to HCV).
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination.
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Safety assessment of new candidate malaria vaccines ChAd63 CS | Participants will be followed for the duration of the study, an expected average of 12 months
  To assess the safety of new candidate malaria vaccines ChAd63 CS administered alone and with MVA CS in a prime-boost regime to healthy volunteers by recording local and systemic solicited and unsolicited adverse events.

SECONDARY OUTCOMES:
Assessment of immune response induced by vaccination | Participants will be followed for the duration of the study, an expected average of 12 months
  To assess the humoral and cellular immune responses generated by ChAd63 CS when administered to healthy volunteers alone and with MVA CS by assessing induced antibody and T cell response to the vaccine insert.

CONTACTS AND LOCATIONS:
Overall Officials: Sam McConkey, Principal Investigator — Clinical Research Centre Royal College of Surgeons in Ireland (RCSI)
Locations (1):
- Clinical Research Centre Royal College of Surgeons in Ireland (RCSI), Beaumont Hospital, Dublin, Ireland

REFERENCES:
- [Derived] de Barra E, Hodgson SH, Ewer KJ, Bliss CM, Hennigan K, Collins A, Berrie E, Lawrie AM, Gilbert SC, Nicosia A, McConkey SJ, Hill AV. A phase Ia study to assess the safety and immunogenicity of new malaria vaccine candidates ChAd63 CS administered alone and with MVA CS. PLoS One. 2014 Dec 18;9(12):e115161. doi: 10.1371/journal.pone.0115161. eCollection 2014. PMID 25522180